CLINICAL TRIAL: NCT03212261
Title: Promoting Resiliency Among Lymphoma Survivors: The 3RP-Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Giselle K. Perez Lougee, Instructor in Psychiatry at Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-063
Record Dates: First submitted 2017-06-21; First posted 2017-07-11 (Actual); Results first posted 2019-10-02 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Lymphoma
Keywords: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3RP-Lymphoma (Experimental): -An adapted version of the 3RP (3RP-Lymphoma) for lymphoma survivors recently completing cancer treatment. The adapted program incorporates the three prongs of the 3RP: RR elicitation, stress awareness, and adaptive strategies. It will be delivered in weekly sessions over the course of approximately 8 weeks.
  Interventions: Behavioral: 3RP-Lymphoma

INTERVENTIONS:
Behavioral: 3RP-Lymphoma — An adapted version of the Relaxation Response Resiliency Program (3RP) for individuals who have recently completed treatment for lymphoma.
  Other Names: Relaxation Response Resiliency Program for Lymphoma

SUMMARY:
The Relaxation Response Resiliency Program (3RP) was developed by researchers at the MGH Benson-Henry Institute for Mind Body Medicine; This program has recently been adapted to target the needs of individuals who have completed treatment for lymphoma (3RP-Lymphoma).

DETAILED DESCRIPTION:
The Relaxation Response Resiliency Program, or 3RP, was developed by researchers at the MGH Benson-Henry Institute for Mind Body Medicine. The 3RP is a group program that-through a variety of mind-body approaches, such as imagery, relaxation, and yoga-seeks to buffer stress and promote psychological resiliency and physical well-being.

The 3RP has not yet been carried out with individuals who have recently completed treatment for lymphoma. As such, the investigators have adapted the standard 3RP program to target the specific needs of lymphoma patients who are transitioning off active treatment. The investigators are conducting this study to see if the adapted program, the 3RP-Lymphoma, is effective at reducing stress and stress-related symptoms for people who have completed treatment for lymphoma within the past two years. To develop the 3RP-Lymphoma, the investigators conducted interviews with patients who had recently completed treatment to learn about their experiences and their preferences for topics they would want to include in a program tailored to their specific needs. The current phase of the feasibility study will examine if the adapted program is feasible, acceptable, and helps promote stress management among lymphoma survivors who are in the early stages of completing cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-64
* Within 2 years post-treatment completion for lymphoma
* English speaking
* Able and willing to provide informed consent
* Cancer treatment or follow-up for lymphoma at the MGH Cancer Center

Exclusion Criteria:

* Unwilling or unable to participate in the study
* Unable to speak or read English
* Is medically, psychiatrically, or otherwise unable to participate (as determined by a physician or study PI)
* Unwilling or unable to participate in group 3RP sessions delivered via the Partners Telehealth videoconferencing software
* Participation in qualitative interview during Phase 1 (DF/HCC 16-396)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giselle K. Perez, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening and recruitment occurred from August through December 2017. There were a few subjects who expressed interest in discussing participation in January 2018 due to the holidays, which led to their enrollment in January 2018. However, the active recruitment period occurred from August through December 2017.
Pre-assignment Details: Individuals who signed consent but who are found to be unable to use the videoconferencing software during the brief test call will be considered ineligible for the study. Two people fell into this category.
Period: Overall Study
Arm/Group | 3RP-Lymphoma
Started | 37 (Enrolled: eligible at time of approach and signed a consent.)
Remained Eligible | 35
Baseline Completion (Eligible patients who completed the baseline survey) | 30 (Lost patients: Technology difficulties (n=2), Family Emergency (n=1), Too busy (n=3), LTFU (n=1))
Program Initiation (4 people completed the baseline survey but did not start the program) | 26 (Lost patients: Tech trouble no first visit (n=1), Too busy/no time (n=2), LTFU (n=1))
Post-intervention Survey (# of people who completed the post-treatment survey (~8 weeks)) | 22 (Lost to follow up (n=4))
One Month Follow-up (# of people who completed the one month follow-up survey (~4 weeks after intervention completion).) | 21 (Lost to follow up (n=1))
Completed | 21
Not Completed | 16
Not completed — Became ineligible d/t tech | 2
Not completed — Tech Trouble- No first study visit | 1
Not completed — Lost to Follow-up | 7
Not completed — Family Emergency | 1
Not completed — Too busy/ No time | 5

BASELINE CHARACTERISTICS:
Population: This number consists of the number of enrolled participants who initiated and completed at least one of the 3RP-lymphoma sessions
Groups:
- 3RP-Lymphoma: Individuals who initiated and participated in any 3RP-lymphoma session
Arm/Group | 3RP-Lymphoma
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.41 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Program Feasibility: Number of Participants Who Completed at Least 75% of the Treatment Sessions
Description: The investigators will evaluate program feasibility by examining rates of treatment completion. Participants who complete at least 75% of the treatment sessions will be identified as treatment completers.
Time Frame: 1 month after completing the 3RP-Lymphoma program
Population: These are people who enrolled and completed at least one 3RP-lymphoma session. This will serve as our denominator to examine the number of people who complete at least 75% of treatment sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | 3RP-Lymphoma
Number analyzed (Participants) | 26
Participants | 20

2. Primary Outcome: Number of Participants Who Found the 3RP Program Acceptable
Description: Acceptability will be assessed at the one-month follow up data collection period with five questions on the 3RP acceptability questionnaire rated on a 4-point Likert scale (1=not at all to 4=very much); higher scores mean higher levels of acceptability.
Time Frame: 1 month after completing the 3RP-Lymphoma program
Measure: Count of Participants; unit: Participants
Groups:
- 3RP-Lymphoma: Individuals who initiated and participated in any 3RP-lymphoma session and completed the 1 month follow up survey
Arm/Group | 3RP-Lymphoma
Number analyzed (Participants) | 21
Participants
  Enjoyable: Somewhat/Very | 21
  Enjoyable: Not at all/Not very | 0
  Helpful: Somewhat/Very | 21
  Helpful: Not at all/Not very | 0
  Relevant: Somewhat/Very | 21
  Relevant: Not at all/Not very | 0
  Convenient: Somewhat/Very | 19
  Convenient: Not at all/Not very | 2
  Somewhat/Very likely to do RR in the future: Somewhat/Very | 21
  Somewhat/Very likely to do RR in the future: Not at all/Not very | 0

3. Secondary Outcome: Number of Participants Who Were Eligible to Provide and Provided Hair Cortisol Samples
Description: The investigators will explore the feasibility and acceptability of collecting hair samples to examine levels of cortisol, a stress biomarker.
Time Frame: 1 month after completing the 3RP-Lymphoma program
Population: Of the 26 participants who participated in the program, only 20 patients were actually able to provide a hair sample. Reasons why they were no longer eligible were because they either had no hair (n=5), or because they reported taking a steroid at the time of collection (n=1).
Measure: Count of Participants; unit: Participants
Arm/Group | 3RP-Lymphoma
Number analyzed (Participants) | 26
Participants
  Total eligible to provide a sample | 20
  Total provided sample based on # eligible: number analyzed (Participants) | 20
  Total provided sample based on # eligible | 14

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from all participants who initiated treatment (N=26). Adverse events were monitored throughout the duration of the intervention, which was approximately 8 weeks for every participant.
Description: None to report
Arm/Group | 3RP-Lymphoma
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/61/NCT03212261/Prot_SAP_000.pdf